CLINICAL TRIAL: NCT00850421
Title: A Single-Center Pharmacoeconomic Pilot Study of BOTOX® (Botulinum Toxin Type A) for the Prophylactic Treatment of Migraine Headaches
Brief Title: Pilot Study of BOTOX for Migraine Headaches
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recently published BOTOX efficacy data and study design deficits.
Sponsor: HealthPartners Institute (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01837-04-C
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Results first posted 2013-09-18 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2013-07

CONDITIONS: Migraine Headache
Keywords: migraine headache; Botulinum Toxin Type A; BOTOX; BTX-A
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botulinum Toxin Type A (Other)
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — 100 Units - Dilution: 25U/ml (4:1 BOTOX/preservative free saline)
  Other Names: BOTOX

SUMMARY:
The purposes of this study are to assess whether subjects treated with BOTOX will:

1. have a decrease in the frequency and intensity of migraine headaches
2. experience improvements in quality of life
3. experience a reduction in the frequency of health care services obtained.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 18 years of age
* Subject has an established history of migraine headache, with or without aura, per IHS criteria (1.2.1 or 1.1), for at least 6 months prior to screening.
* Subject receives primary health care from Park Nicollet Health Services.

Exclusion Criteria:

* Subject has received previous injections of botulinum toxin of any serotype for any reason, within the 6 months prior to study participation.

Additional eligibility will be discussed at point of contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Taylor, MD, Principal Investigator — Park Nicollet Health Services
Locations (1):
- Park Nicollet Health Services, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A
Started | 35
Completed | 18
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: To Determine Whether Resource Utilization is Decreased in Subjects Treated With BOTOX Injections for Episodic Migraine Headache.
Time Frame: 190 days
Population: Mid-enrollment statistical review determined study should not continue, due to recently published BOTOX efficacy data and study design deficits. Not possible to summarize as PI left the institution and did not provide location of the data
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 0

2. Secondary Outcome: To Determine Whether Quality of Life is Improved in Subjects Treated With BOTOX Injections for Episodic Migraine Headache.
Time Frame: 190 days
Population: as for outcome 1
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 0

3. Secondary Outcome: To Assess the Effect of BOTX Injections on the Frequency and Intensity of Migraine Episodes in Subjects With Episodic Migraine Headache.
Time Frame: 190 days
Population: as for outcome 1
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin Type A
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 6/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=35)
Sore throat (Infections and infestations) | 2
Soreness, posterior neck (Musculoskeletal and connective tissue disorders) | 2
Urinary tract infection (Renal and urinary disorders) | 2

LIMITATIONS AND CAVEATS:
This study was terminated and PI left organization. No results available to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes